CLINICAL TRIAL: NCT05462054
Title: A Phase 0 Non-interventional, Multi-center, Natural History Study in Pediatric Patients with Syntaxin Binding Protein 1 (STXBP1) Encephalopathy with Epilepsy
Brief Title: Natural History Study in Pediatric Patients with STXBP1 Encephalopathy with Epilepsy
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawn, no patients enrolled
Sponsor: Capsida Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CAP-002-501
Record Dates: First submitted 2022-07-05; First posted 2022-07-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: STXBP1 Encephalopathy with Epilepsy
Keywords: STXBP1; Epilepsy; Seizures; Epileptic encephalopathy; Genetic Diseases, Inborn
MeSH Terms: conditions — Epileptic Encephalopathy, Early Infantile, 4; Epilepsy; Seizures; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — STXBP1 gene mutation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective, non-interventional, longitudinal study designed to characterize the natural history of STXBP1 related encephalopathy with epilepsy, in participants ≤ <5 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, > 1 day to ≤ 5 years of age at the time of informed consent.
* Diagnosed with seizure disorder
* Presence of a STXBP1 gene mutation. Historical documentation is sufficient to support eligibility for the study. Confirmatory testing will be obtained at baseline and performed by a CLIA certified laboratory
* Written informed consent provided by a parent or legal guardian

Exclusion Criteria:

* History of prior gene therapy treatment
* Current enrollment in an interventional study or has received an investigational drug within 30 days or fewer than 5 half-lives prior to screening visit, whichever is longer
* Treatment with any antisense oligonucleotide therapy within 6 months prior to screening and anticipate remaining on treatment throughout the study
* The presence of a confirmed mutation in a gene other than STXPB1 that is known to contribute to a neurodevelopmental disability
* Presence of a significant non-STXBP1 related central nervous impairment/behavioral disturbance that would confound the scientific rigor or interpretation of results of the study
* History of prematurity (defined as gestational age <35 weeks), interventricular hemorrhage, structural brain deficit or congenital heart disease
* Requires mechanical ventilation or non-invasive respiratory support such as continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BiPAP) at the time of informed consent

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: ≤5 years of age with STXBP1 related encephalopathy with epilepsy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Changes in neurodevelopmental parameters of adaptive behavior function over time utilizing the Vineland Adaptive Behavior Scales-II (VABS-II) Age-equivalent Scores | 2 Years
  The Vineland Adaptive Behavior Scales, Second Edition (Survey Interview Form) is a measure of adaptive behavior in children, adolescents and adults. It yields an overall standard score (Adaptive Behavior Composite, ABC) and age standard scores in four domains. ABC scores have a mean of 100 and a standard deviation of 15 (range = 20 to 160). Higher scores suggest a higher level of adaptive functioning.
Changes in neurodevelopment parameters over time utilizing an age appropriate assessment. | 2 Years
  The determination of whether a patient received Bayley Scales of Infant Development-III (BSID-III) is based on an algorithm that includes the patient's calendar age and VABS-II age-equivalent score (See Outcome 1). The BSID-III is a series of measurements to assess the motor (fine and gross), language (receptive and expressive), and cognitive development of infants and toddlers and consists of a series of developmental play tasks. contains two scoring systems of composite scores and percentile ranks. The normal range for composite scores is between 40-160 with mean at 100 and 0-99 for the percentile ranks. Higher scores mean a better outcome.
Changes in neurodevelopment parameters over time utilizing an age appropriate assessment. | 2 Years
  The determination of whether a patient received Kaufman Assessment Battery for Children-II (KABC-II) is based on an algorithm that includes the patient's calendar age and VABS-II age-equivalent score (See Outcome 1). The KABC-II is an individually administered measure of processing and reasoning abilities. The scoring range is 69 and below through 131 or greater. Higher scores mean a better outcome.
Changes in seizure frequency over time | 2 Years
  Seizure diary

SECONDARY OUTCOMES:
Changes in communication ability over time | 2 Years
  Observer-Reported Communication Ability (ORCA) Outcome Measure. The ORCA measure produces a single score that is an estimate of an individual's overall level of communication ability. Higher ORCA scores reflect greater communication ability; the mastery of expressive, receptive, and pragmatic types of communication and higher vocabularies for verbal words and symbols on assistive devices. The ORCA T-score range is from 26.82 to 83.24.
Changes in sleep behavior over time | 2 Years
  Patient sleep habits will be assessed using Children's Sleep Habits Questionnaires (CSHQ).
Changes in electroencephalogram (EEG) recording over time | 2 Years
  Standard EEG, lasting approximately 1 hour, to assess the presence of epileptiform activity.
Changes in motor function over time utilizing an age appropriate assessment. | 2 Years
  The Hammersmith Infant Neurological Examination (HINE) is aimed to be used for infants between 3 and 24 months of age and assess different aspects of neurological function: cranial nerve function, movements, reflexes and protective reactions and behavior, as well as some age-dependent items that reflect the development of gross and fine motor function. Each item is scored 0-3, higher scores mean a better outcome.
Changes in motor function over time utilizing an age appropriate assessment. | 2 Years
  The Gross Motor Function Measure-88 is aimed to be used for children 5 months or older of age and assess changes in gross motor function over time. Each item is scored 0-3, higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Capsida Biotherapeutics, Inc.

IPD SHARING:
Plan to Share IPD: Undecided